CLINICAL TRIAL: NCT01744132
Title: Overcoming Barriers in Vision Care Utilization of African Americans With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Alabama at Birmingham (Other); University of Miami (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Julia Haller, Prinipal Investigator, Ophthalmologist-in-Chief, Wills Eye
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U58DP002655 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetic Retinopathy; Diabetes Mellitus
Keywords: eye care utilization; ophthalmology; educational intervention; public health screening
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aim 3: Contract (Experimental): Half of patients screened in the pharmacy are selected to a contract group, which encourages patients to review the results of the screen, share the results with their PCP, and schedule and attend a follow-up appointment with an ophthalmologist if the results are abnormal.
  Interventions: Behavioral: Aim 3: Contract
- Aim 3: Control (No Intervention): No contract is signed for half of the patients screened in Aim 3.

INTERVENTIONS:
Behavioral: Aim 3: Contract
  Arms: Aim 3: Contract

SUMMARY:
The goal of this project is to implement a Collaborative Translational Research Center (TRC) Network Study which aims to assure optimal two-way communication between ophthalmologists and their patients' primary care physicians (PCP). The Collaborative TRC Network Study will have 2 objectives:

* To design and develop common research protocols to develop a 4-year retrospective database (2007-2010) that compiles electronic billing and medical chart information that can be used to study individual-level, clinical-level and system-level factors that impact access to and quality of vision care;
* To evaluate adherence to dilated fundus exams (DFEs) follow-up as the primary measureable quality indicator, and its relationship to the patients' demographics, ethnicity, socioeconomic status (SES), severity of diabetic retinopathy (DR), other ocular and medical co-morbidities, presence of HA1C, and primary care provider (PCP) communication.

By enhancing communication and strengthening the clinical information exchanged between PCPs and eye care professionals, this Collaborative TRC Network study will help to overcome barriers to obtaining ongoing DFEs and reduce disparities in vision care utilization.

DETAILED DESCRIPTION:
Since its inception in October 2010 Collaborative Network Research Study at the Wills Eye Institute has aimed:

1. to establish a retrospective analysis of existing ophthalmic data sets to assess and evaluate system-level and individual-level factors that impact access to and quality of vision care in patients with diabetes;
2. to implement telephone-based and educational interventions to improve DFE follow-up adherence in African Americans with diabetes utilizing a prospective, cluster-based, randomized cohort design;
3. to determine the feasibility and effectiveness of using a non-invasive, non-mydriatic fundus camera (Nidek) in a community-based pharmacy setting to screen and detect diabetic retinopathy and other ocular diseases among individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria for Aim 1:

1. Age ≥ 18 years
2. Type 2 diabetes mellitus
3. Had a dilated fundus exam (DFE) within the past four years (2007-2010).

Exclusion Criteria for Aim 1:

1) Pregnant women

Inclusion Criteria for Aim 2 and 3:

1. Age ≥ 18 years
2. Type 2 diabetes mellitus
3. Access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
All Aims: DFE follow-up adherence rate | 2 years
  In Aim 1 and Aim 2 specifically the influence patients' ethnicity and severity of diabetic retinopathy will be examined with the rate of dilated fundus examine (DFE) follow-up adherence.
  In Aim 3, the rate of DFE follow-up adherence will be examined for both patients in the contract and the no contract group.

SECONDARY OUTCOMES:
Aim 3: Rates of ocular disease | 2 years
  In Aim 3, the occurrence of diabetic retinopathy, glaucoma, cataracts, and other ocular diseases will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Haller, Principal Investigator — Wills Eye Hospital
Locations (1):
- Jefferson Pharmacy, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keenum Z, McGwin G Jr, Witherspoon CD, Haller JA, Clark ME, Owsley C. Patients' Adherence to Recommended Follow-up Eye Care After Diabetic Retinopathy Screening in a Publicly Funded County Clinic and Factors Associated With Follow-up Eye Care Use. JAMA Ophthalmol. 2016 Nov 1;134(11):1221-1228. doi: 10.1001/jamaophthalmol.2016.3081. PMID 27632231
- [Background] Murchison AP, Friedman DS, Gower EW, Haller JA, Lam BL, Lee DJ, McGwin G Jr, Owsley C, Saaddine J, Insight Study Group. A Multi-Center Diabetes Eye Screening Study in Community Settings: Study Design and Methodology. Ophthalmic Epidemiol. 2016;23(2):109-15. doi: 10.3109/09286586.2015.1099682. Epub 2016 Mar 7. PMID 26949832
- [Background] Callinan CE, Kenney B, Hark LA, Murchison AP, Dai Y, Leiby BE, Mayro EL, Bilson J, Haller JA. Improving Follow-Up Adherence in a Primary Eye Care Setting. Am J Med Qual. 2017 Jan/Feb;32(1):73-79. doi: 10.1177/1062860615616860. Epub 2016 Jul 10. PMID 26656245
- [Background] Aleo CL, Murchison AP, Dai Y, Hark LA, Mayro EL, Collymore B, Haller JA. Improving eye care follow-up adherence in diabetic patients with ocular abnormalities: the effectiveness of patient contracts in a free, pharmacy-based eye screening. Public Health. 2015 Jul;129(7):996-9. doi: 10.1016/j.puhe.2015.05.012. Epub 2015 Jun 25. PMID 26119987
- [Background] Storey PP, Murchison AP, Pizzi LT, Hark LA, Dai Y, Leiby BE, Haller JA. IMPACT OF PHYSICIAN COMMUNICATION ON DIABETIC EYE EXAMINATION ADHERENCE: Results From a Retrospective Cohort Analysis. Retina. 2016 Jan;36(1):20-7. doi: 10.1097/IAE.0000000000000652. PMID 26098386